CLINICAL TRIAL: NCT03218150
Title: Cranioplasty: Autogenous Bone Graft Versus Artificial Substitutes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaeddin Mohamed Ali, resident doctor, Assiut University
Other Study IDs: Assiut cranioplasty
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Cerebral Decompression Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- bone cement group: patient underwent to cranioplasty reconstruction with customized hydroxyapatite prosthesis
  Interventions: Procedure: cranioplasty
- titanium mesh group: patient underwent to cranioplasty reconstruction with titanium mesh
  Interventions: Procedure: cranioplasty
- autologous bone group: patient underwent to cranioplasty reconstruction with autologous bone graft
  Interventions: Procedure: cranioplasty

INTERVENTIONS:
Procedure: cranioplasty — . The margins of the craniectomy defects exposed, and the bone flaps fixed in their original positions using wires or titanium plates with screws. As prophylaxis, all patients intravenously administered with pre- and postoperative antibiotics.
  In cases of artificial substitutes , The polymethyemethacrylate implant fixed to the defective region with titanium plates and self-tapping screws.

SUMMARY:
Prospective, comparative, observational study.

The project's aim is long term follow up of patient's having skull bone defects due to traumatic or lesion resection causes, treated , in standard clinical practice, with autologous bone graft , bone cement or titanium mesh and to compare the clinical outcome and safety among the 3 types of treatment.

Eligibility to each treatment will respect the standard clinical practice.

Primary outcome: minimize post operative infection

Secondary outcomes: decrease operation time , clinical and psychological improvement of the patient, decrease the cost on the patient

DETAILED DESCRIPTION:
Cranioplasty is the surgical intervention to repair cranial defects. The aim of cranioplasty is not only a cosmetic issue; also, the repair of cranial defects gives relief to psychological drawbacks and increases the social performances. Many different types of materials were used throughout the history of cranioplasty. With the evolving biomedical technology, new materials are available to be used by the surgeons. Although many different materials and techniques had been described, ongoing researches on both biologic and non biologic substitutions continue aiming to develop the ideal reconstruction material.

Autologous bone grafts remain the best option for adult and pediatric patients with viable donor sites and small-to-medium defects. Large defects in the adult population can be reconstructed with titanium mesh and polymethylmethacrylate overlay with or without the use of computer-assisted design and manufacturing customization. Advances in alloplastic materials and custom manufacturing of implants will have an important influence on cranioplasty techniques in the years to come.

ELIGIBILITY:
Inclusion Criteria:

1. All patients that have reconstructive surgery of cranial defects due to traumatic or lesion resection causes .
2. Age older than 10 and less than 60 years
3. Provided written informed consent

Exclusion Criteria:

1. Cases of cranial defects due to congenital anomalies or growing skull fractures .
2. Severe disease with limited life expectancy of less than one year

Ages: 10 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient's that need cranioplasty surgery admitted in assiut university hospital
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
safety : minimize incidence of infection | 360 days after surgery
  incidence of adverse events ((infection, reabsorption))

SECONDARY OUTCOMES:
efficacy | 60 , 120 , 360 days after surgery
  quality of life improvement evaluation : (( glasgow coma score))

IPD SHARING:
Plan to Share IPD: No